CLINICAL TRIAL: NCT00377065
Title: Early Access of MK0518 in Combination With an Optimized Background Antiretroviral Therapy (OBT) in Highly Treatment Experienced HIV-1 Infected Patients With Limited to No Treatment Options
Brief Title: Early Access of MK0518 in Combination With an Optimized Background Antiretroviral Therapy (0518-023)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0518-023; MK0518-023; 2006_031
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

INTERVENTIONS:
Drug: raltegravir — raltegravir 400 mg P.O. bid tablet twice daily for 12 weeks
  Other Names: MK0518; ISENTRESS™

SUMMARY:
This is a treatment use study to provide early access to MK0518 for the treatment of HIV-1 infection in patients who have limited or no treatment options due to virological failure, resistance, or intolerance to multiple antiretroviral regimens. Enrollment in this study is patient driven. Investigators are not proactively assigned. There is no target sample size and duration of the study is indefinite. For information on how to enroll in the study, see link below.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patients who have limited or no treatment options and have documented resistance

Exclusion Criteria:

* Patient has previously been on MK0518 therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC